CLINICAL TRIAL: NCT01447810
Title: Constraint Induced Movement Therapy in a Pediatric Oncology Population (SJCIT): A Pilot Study
Brief Title: Constraint-Induced Movement Therapy in a Pediatric Oncology Population
Acronym: SJCIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SJCIT
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2014-09

CONDITIONS: Hemiplegia; Brain Tumor
Keywords: Constraint-Induced Movement therapy; Pediatric; Hemiplegia; Brain Tumor; Rehabilitation
MeSH Terms: conditions — Hemiplegia; Brain Neoplasms | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Other: Focused rigidity bi-valve long arm cast

INTERVENTIONS:
Other: Focused rigidity bi-valve long arm cast — Two focused rigidity bi-valve long arm (upper arm to finger tips) casts will be fabricated for each participant on day one of the constraint-induced therapy (CIT) program. Focused rigidity casting materials are water proof and latex/fiberglass free. Focused rigidity casting does not require use of a cast saw for removal thus decreasing potential for anxiety during the casting process. Casts will be fabricated by therapist trained in the casting technique.
  Other Names: constraint-induced therapy

SUMMARY:
Hemiplegia (weakness or poor muscle function on one side of the body) is a neurological impairment which can occur in children as a result of a brain tumor or related treatment. This impairment can negatively impact the child's functional abilities and movement development, making it difficult for them to play, learn to feed, dress or bathe themselves, and to participate fully in home, daycare, or school environments. Poor movement skills may also impact overall quality of life. Constraint Induced Therapy is a rehabilitation technique which has been found to improve the child's abilities to move their arms following neurological injuries like stroke and traumatic brain injury in both adults and children.

The aim of this study is to evaluate the feasibility of implementing a constraint induced movement therapy program in a small group of children with a brain tumor and hemiplegia. Children who participate in the program may experience improved ability to use their weak arm leading to increased participation in meaningful activity and improved quality of life.

DETAILED DESCRIPTION:
Constraint Induced Therapy (CI Therapy) is based on the theory of "learned non-use." Following an event that impacts the brain (stroke, brain injury etc.), the messages from the brain to the arm and the messages from the arm to the brain are interrupted in the area of the brain where the injury occurred and in a small surrounding area. The arm is often inefficient and difficult to use. Over time, even after swelling in the brain decreases, movement of the affected arm continues to be more effortful and the child becomes quite accustomed to completing activities with the unaffected arm only. Additionally, because the child has not used the weak arm for a while, the part of the brain that is ready to receive signals and give commands to the arm or leg is "quiet" and does not work like it used to. The theory of "learned no-nuse" has lead to the development of the CI Therapy approach which is comprised of the following principles:

* Constraint - the strong or normal arm/leg is restrained, forcing use of the weaker arm/leg during treatment.
* Practiced Use - the weak limb is treated by engaging the child in structured practice of specific movements and functional skills.
* Transfer Package - a home program is developed for the child to use with his or her caregivers that focuses on facilitating carryover of learned skills into the real world environment.

This theory hypothesizes that, because the nervous system, particularly in the child, has plasticity (can be shaped and learn to do new things), CI Therapy will facilitate cortical (brain) reorganization, and help the child overcome learned non-use, eventually leading to improved function of the weak arm or leg.

Phase 1: Initial evaluations will be completed on day 1 of the program. They include interview questions and direct assessment of the participant's ability to use the affected arm as well as to participate in meaningful age-appropriate activities. These assessments include the Motor Activity Log, The Pediatric Arm Function Test, the Inventory of New Motor Activities and Programs, the Pediatric Quality of Life Inventory, and the Preschool Activity Card Sort or Children's Assessment of Activity Preferences.

Phase 2: The participant completes an intensive occupational therapy program which consists of 15 three-hour therapy sessions (5 days per week for 3 weeks). Throughout the three week program the un-involved arm will be constrained with a removable cast. The cast is to be worn 24 hours per day throughout the 3 week program with the exception of regularly scheduled cast changes, washings and skin checks completed by the treating occupational therapist. During the direct intervention sessions, a focus of therapy is on facilitation of new motor skills for the affected arm. Play is utilized as a means to motivate the pediatric participants with activities and exercises specifically chosen to facilitate new motor skills. The program also includes a variety of tools and activities caregivers will complete increasing adherence to the program outside of the direct intervention sessions and to facilitate transfer of affected upper extremity use into the real world environment.

Phase 3: Immediately following the 3 week intervention program the participant's performance is re-assessed. Additionally weekly follow up evaluations are completed by phone for a period of one month. Three months following the intervention program the participant will return for follow up evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed hemiplegia of an upper extremity as documented by physician or rehabilitation clinician in the medical record
* Diagnosis of brain tumor
* English speaking
* Participant has demonstrated the ability in the past to move the elbow >70 degrees and has some purposeful movement in the hand (ability to initiate a gross grasp).
* Parent/legal guardian is willing to give consent to participate in the study.
* Child is willing to give assent in the study if seven years old or older.

Exclusion Criteria:

* Severe hemiplegia and resulting active range of motion deficits at the affected upper extremity as defined by the following:

  * < 30 degrees active shoulder flexion or abduction
  * Inability to initiate active elbow flexion or extension.
  * Inability to initiate movements at the of wrist, finger or thumb
* Uncontrolled seizures that interfere with daily activities, as this would interfere with the participant's ability to fully participate in the CI Therapy program.
* Pain that significantly interferes with the participant's ability to fully participate in the intensive therapy program. This includes pain related to subluxation of the shoulder, as measured by a pain rating of 5/10 or greater on the FACES or Numeric Pain Scale.
* Currently receiving oral or intravenous chemotherapy or radiation therapy.
* Inability or unwillingness of legal guardian to give written informed consent.
* Child is unwilling to give assent if seven years old or older.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of participants who complete the study. | One (1) year
  To evaluate the feasibility of conducting a 3-week constraint-induced therapy program in patients with upper extremity hemiplegia as a result of a tumor. We will conclude that conducting this constraint induced therapy program is not feasible if more than 2 patients out of eight patients do not complete the program for any reason, with exception those outlined as excused reasons for absence from a therapy sessions (acute illness of the participant, illness of a parent, or other interruptions considered allowable/unavoidable by the study PI).

SECONDARY OUTCOMES:
Frequency of extremity use. | Baseline, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 4 months
  To describe the change in amount of extremity use at pre-intervention, post-intervention and at follow-up.
Quality of extremity function. | Baseline, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 4 months
  To describe the change in quality of extremity use at pre-intervention, post-intervention and at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Sparrow, OTD, OTR/L, Study Chair — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols